CLINICAL TRIAL: NCT05068908
Title: Brain Connectivity Patterns in Chronic Temporomandibular Joint Disorders
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: DENT-2020-29282
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Temporomandibular Joint Disorders; Temporomandibular Joint Pain
MeSH Terms: conditions — Chronic Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low-impact chronic painful temporomandibular disorder (TMD) cases: Participants whose chronic painful TMD is determined to be low-impact. Visits include a standardized clinical examination using the Diagnostic Criteria for TMD (DC/TMD) protocol, psychosocial questionnaires completion, sensory and endogenous pain modulation (EPM) testing and a multi-modal Magnetic Resonance Imaging (MRI) data acquisition.
- High- impact chronic painful temporomandibular disorder (TMD) cases: Participants whose chronic painful TMD is determined to be high-impact. Visits include a standardized clinical examination using the Diagnostic Criteria for TMD (DC/TMD) protocol, psychosocial questionnaires completion, sensory and endogenous pain modulation (EPM) testing and a multi-modal Magnetic Resonance Imaging (MRI) data acquisition.
- Pain-free controls: Participants without chronic painful TMD. Visits include a standardized clinical examination using the Diagnostic Criteria for TMD (DC/TMD) protocol, psychosocial questionnaires completion, sensory and endogenous pain modulation (EPM) testing and a multi-modal Magnetic Resonance Imaging (MRI) data acquisition.
- Pilot study-MRI optimization group: A pilot study will be conducted separately from the "main project" for optimization of MRI parameters, where up to five participants will be recruited as a separate group to undergo only MRI sessions (single study visit). The goal is to optimize the parameters of the main project's MR imaging protocol in order to minimize imaging distortions related to the presence of the thermodes in close proximity to the field of view for the brain.

SUMMARY:
This study addresses the timely problem of painful temporomandibular disorders (TMD), the most common cause of orofacial pain second only to tooth pain. Findings from previous studies suggest that dysregulation of connectivity within specific brain circuits is part of chronic pain pathophysiology. This study will identify connectivity patterns within those brain circuits as potential signatures for pain- related disability in chronic TMD pain participants. New knowledge regarding these brain connectivity patterns is expected to be significant because it will support improved phenotyping of this heterogeneous participant population. It is also expected that this finding can potentially be extrapolated to other chronic pain conditions, such as back pain, migraine headache, and fibromyalgia that are frequently comorbid conditions in chronic TMD participants.

DETAILED DESCRIPTION:
Evidence of dysregulation of brain circuits in chronic pain in general and in chronic temporomandibular disorder (TMD) pain specifically is well documented. Among putative brain circuits involved in chronic pain pathophysiology are thalamocortical brain pathways, which transmit nociceptive signals centrally from peripheral tissues. Pathways between the medial prefrontal cortex (mPFC) and the periaqueductal gray (PAG) are considered part of an antinociceptive brain circuit, since they are necessary to engage endogenous pain modulation. Dysfunction of endogenous pain modulation has been systematically reported in chronic pain patients, and a meta-analysis of clinical studies of TMD patients done by the Principal investigator and others showed increased pain facilitation and impaired pain inhibition in patients relative to pain-free controls.

Endogenous pain modulation can be assessed by psychophysical methods. For instance, pain facilitation can be assessed with temporal summation of pain (TSP) using brief noxious stimuli presented repeatedly over peripheral tissues at >0.3 Hz. Pain inhibition can be assessed with conditioned pain modulation (CPM) by presenting noxious stimuli over a body site during concurrent noxious stimuli elsewhere to induce pain inhibition. Neuroimaging studies in pain-free controls showed that functional connectivity within thalamocortical and antinociceptive brain circuits are related to increased TSP and reduced CPM responses, respectively. It is unknown if connectivity patterns within the thalamocortical and antinociceptive brain circuits are altered in chronic TMD patients, reflecting endogenous pain modulation dysfunction. Corticolimbic pathways connecting the mPFC, amygdala and nucleus accumbens are thought to play a key role in chronic pain and specifically, in emotion-driven modulation of nociceptive signals. Recently a longitudinal study showed that functional and structural connectivity patterns determined from neuroimaging data between these regions predict transition from acute to chronic back pain. A population study of TMD pain patients showed that approximately 64% of these patients also present with comorbid low back pain, thus it is possible that chronic TMD pain patients may display brain connectivity patterns that are similar to those identified in persistent back pain patients.

Functional brain connectivity is usually assessed from resting-state functional magnetic resonance imaging (fMRI), where participants lay at rest during fMRI scans to measure intrinsic functional connectivity (FC). Connectivity patterns within the thalamocortical, corticolimbic and antinociceptive circuits described above were determined using this traditional approach for FC assessment. Recent studies departed from this traditional approach and assessed FC during presentation of noxious stimuli during fMRI data acquisition and identified evoked FC changes. These studies' results suggest that noxious stimuli affect connectivity patterns in brain circuits involved in pain processing in pain-free participants and in fibromyalgia patients. Thus, it is reasonable that psychophysical testing for pain facilitation (e.g., TSP) and pain inhibition (e.g., CPM) could reflect changes in connectivity patterns within brain circuits associated with pain modulation. If confirmed, these evoked connectivity patterns identified from engaging endogenous pain modulation could serve as a "signature" for pain modulation in individuals, similar to a "functional connectome fingerprinting" demonstrated to predict fluid intelligence in healthy participants using data from the Human Connectome Project (HCP).

Taken together these results suggest new approaches to investigate dysregulation of brain circuits in chronic TMD pain with a focus on brain connectivity, that can serve as unique chronic pain "signatures" related to endogenous pain modulation function. There is a critical need to determine the potential of brain circuits' connectivity patterns to serve as signatures for pain- related disability. Addressing this critical need will provide novel ways to identify subgroups of chronic TMD pain patients who respond poorly to treatment. Closing this gap in our knowledge has reasonable potential to provide the opportunity for development of precise and valid brain imaging methods supporting refined phenotyping of chronic TMD pain patients leading to early identification of patients with poor prognosis.

Chronic pain causes suffering to more Americans than heart disease, diabetes and cancer combined, and TMD is the second most commonly occurring musculoskeletal condition resulting in pain and disability after chronic back pain. TMD affects approximately 5-12% of the population, with annual estimates of economic impact ranging between $4 billion per the NIDCR and $32 billion according to a study sponsored by the Agency for Healthcare Research and Quality . Pain-related disability significantly impacts patient's quality of life, and a subgroup of chronic TMD pain patients present with high pain-related disability, as identified by the Graded Chronic Pain Scale (GCPS), and these patients have poor prognoses - even with treatment - and greater health care costs.

About half to two-thirds of individuals with TMD seek treatment, and of those approximately 15% will develop chronic pain. Chronic TMD pain patients present with pain persisting ≥6 months, and it is well accepted that chronic TMD pain pathophysiology includes dysregulation of brain circuits. Recent evidence suggests that brain functional and anatomical characteristics, namely connectivity patterns within specific brain circuits, are related to processing, modulation and persistence of pain. Brain connectivity patterns within the thalamocortical circuit are associated with expression of endogenous pain facilitation, while connectivity patterns between prefrontal cortex and brainstem nuclei, an antinociceptive circuit, are related to endogenous pain inhibition. In addition, brain connectivity patterns within corticolimbic pathways involved in the emotion-driven modulation of nociceptive signals predict transition from acute to chronic back pain. These connectivity patterns within thalamocortical, antinociceptive, and corticolimbic brain circuits have not been described in chronic TMD patients, and it is unknown if connectivity patterns within these brain circuits can distinguish chronic TMD patients based on pain-related disability.

ELIGIBILITY:
Inclusion Criteria: Main project

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of study participation.
* All participants will be females (biological sex by self-report) between ages 18 to 65 years (inclusive), as this includes the majority of the patient population at risk for chronic TMD pain.
* Cases and controls will be matched for age within ±3 years, and all participants must be able to understand commands in English to follow study procedures (e.g., during sensory testing).

Pain-free controls

* TMD-Pain screener score less than 3 out of 7 (Screener available as part of the DC/TMD)
* No previous diagnosis for the most common pain-related TMD as defined in the DC/TMD criteria (myalgia, arthralgia, headache attributed to TMD)
* No significant orofacial pain (jaw pain, TMJ pain) in past 3 months ("significant" meaning 5 or more days in any month or any pain during the past month)
* No report of significant pain in the last 3 months elsewhere in the body ("significant" meaning 5 or more days in any month or any pain during the past month), e.g., low back pain, fibromyalgia, migraine headaches
* Not meeting any of the most common pain-related TMD diagnosis as described in the DC/TMD criteria (myalgia, arthralgia, headache attributed to TMD) upon clinical examination following the DC/TMD protocol

Chronic painful TMD cases

* TMD-pain screener score equal to or greater than 3
* Primary TMD caseness criteria: myalgia (masticatory muscle pain) based on clinical exam following the DC/TMD protocol

  * Concurrent arthralgia (TMJ pain) and/or headache attributed to TMD allowed
* Myofascial pain must meet the following criteria:

  * Onset >3 months, occurring >15 days/month on average for >3 months
  * Minimum 10 jaw pain episodes since onset, each episode lasting at least 30 minutes and no less than 2 hours within the day, OR unremitting
* Low-impact TMD pain cases: Graded Chronic Pain Scale (GCPS) grade IIa or lower
* High-impact TMD pain cases: GCPS grade IIb or greater

Inclusion criteria: Patients in MRI Optimization group

* Be age 18-65 (inclusive)
* Provide a signed and dated informed consent form.
* Be willing to comply with all study procedures and be available for the duration of study participation.
* Be able to understand commands in English to follow study procedures.

Exclusion Criteria: Main project

* Traumatic facial injury or surgery on the face/jaw, arms or hands
* Presence of pain related to dental or periodontal pathology
* Currently undergoing active orthodontic treatment
* Pregnant or nursing
* Has any of the following medical conditions by self-report:

  * Renal failure or dialysis
  * Heart disease (examples: uncontrolled arrhythmia or hypertension, cardiomyopathy) or heart failure
  * Non-allergic bronchospasm (chronic obstructive pulmonary disease and emphysema)
  * Diabetes (Type I or II) that is not controlled with medication or diet
  * Hyperthyroidism
  * Uncontrolled seizures
* Used any injection therapy (i.e. tender or trigger point injections, steroid injections), acupuncture, biofeedback, or TENS for the management of facial pain within 2 weeks prior to the screening assessment

  * If undergoing botulinum toxin injections in the head and neck areas, must be 3 months since last set of injections and refrain from this treatment until study has ended
* History of major depression or other major psychiatric disorder requiring hospitalization within the last 6 months prior to the screening assessments
* History of treatment for drug or alcohol abuse within the last 12 months
* Current pain medication use (e.g. opioids, ibuprofen, acetaminophen) that cannot be stopped <24 hours prior to each study visit
* Other conditions/diseases associated with altered pain perception: neurological or developmental disorders (dementia, autism spectrum disorder), neoplasm, multiple sclerosis, trigeminal neuralgia
* MRA contraindications including claustrophobia
* GCPS grade assigned at Visit 1 that does not match grade from screening GCPS (low-, high-impact pain) and it is not possible to assign the potential participant to the correct final group, due to the latter having met their recruitment quota
* Strictly left-handedness by self-report
* Thermal threshold for Pain-50 (determined at Visit 1) is outside the temperature range of 40-49 degrees Celsius
* Lack of access to electronic device with internet connection during the study
* Inability or unwillingness to receive daily text messages during the study
* Inability to complete at least four daily ratings between the Informed consent, Pre- visit 1 procedures and in-person visit 1
* Anything that would place the individual at increased risk or preclude the individual's full compliance with study procedures or completion of the study.

Exclusion criteria: MRI Optimization group

Pregnant or nursing;

* MRI contraindications including claustrophobia;
* Adults lacking capacity to provide informed consent for themselves;
* Unable to understand instructions for sensory testing in English;
* Anything that would place the individual at increased risk or preclude the individual's full compliance with study procedures or completion of the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Visits include a standardized clinical examination using the Diagnostic Criteria for TMD (DC/TMD) protocol, psychosocial questionnaires completion, quantitative sensory testing (QST) using a standard protocol, endogenous pain modulation (EPM) testing and a multi-modal Magnetic Resonance Imaging (MRI) data acquisition.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity (FC) for the thalamocortical brain circuit | 2.5 hours
  Multi-modal MRI data will be used to assess functional connectivity patterns within the thalamocortical brain circuit in chronic TMD pain participants and pain free controls. Functional connectivity will be reported as a unitless value. Neuroimaging will be conducted during Visit 3.
Functional connectivity (FC) for the antinociceptive brain circuit | 2.5 hours
  Multi-modal MRI data will be used to assess functional connectivity patterns within the antinociceptive brain circuit in chronic TMD pain participants and pain free controls. Functional connectivity will be reported as a unitless value. Neuroimaging will be conducted during Visit 3.
Functional connectivity (FC) for the corticolimbic brain circuit | 2.5 hours
  Multi-modal MRI data will be used to assess functional connectivity patterns within the corticolimbic brain circuit in chronic TMD pain participants and pain free controls. Functional connectivity will be reported as a unitless value. Neuroimaging will be conducted during Visit 3.
Anatomical connectivity (AC) for the thalamocortical brain circuit | 2.5 hours
  Multi-modal MRI data will be used to assess anatomical connectivity patterns within the thalamocortical brain circuit in chronic TMD pain participants and pain free controls. Anatomical connectivity will be reported as a unitless value. Neuroimaging will be conducted during Visit 3.
Anatomical connectivity (AC) for the antinociceptive brain circuit | 2.5 hours
  Multi-modal MRI data will be used to assess anatomical connectivity patterns within the antinociceptive brain circuit in chronic TMD pain participants and pain free controls. Anatomical connectivity will be reported as a unitless value. Neuroimaging will be conducted during Visit 3.
Change in anatomical connectivity of corticolimbic brain circuit | 2.5 hours
  Multi-modal MRI data will be used to assess anatomical connectivity patterns within the corticolimbic brain circuit in chronic TMD pain participants and pain free controls. Anatomical connectivity will be reported as a unitless value. Neuroimaging will be conducted during Visit 3.

SECONDARY OUTCOMES:
Temporal Summation of Pain (TSP) and Conditioned Pain Modulation (CPM) responses | 3.5 hours
  To assess correlations between functional connectivity and anatomical connectivity matrices and individual endogenous pain modulation responses, TSP and CPM testing will be conducted. TSP testing uses a thermal device and custom pressure algometers to deliver a single stimulus perceived as "slightly painful" by the participant, followed by 5- or 10-stimuli series repeated at 1 Hz. CPM testing uses a pressure algometer as test stimulus to deliver increasing pressure (50kPa/s rate) to the test site until the participant presses a switch signaling when the pressure sensation first becomes painful. The conditioning stimulus (CS) used to elicit pain inhibition for CPM testing is tonic noxious contact heat applied to the non-dominant volar forearm. CPM testing is also done in triplicate on two occasions: at baseline and during CS applied to the forearm. TSP and CPM responses will be assessed during Visit 2 of the study and reported as percentage values.

CONTACTS AND LOCATIONS:
Overall Officials: Estephan J Moana-Filho, DDS, MS, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States